CLINICAL TRIAL: NCT04019730
Title: The Effect of a Ketogenic Diet on the Exercise Induced Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL6540408118
Record Dates: First submitted 2018-07-06; First posted 2019-07-15 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-07

CONDITIONS: Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low carbohydrate diet (Experimental): less than 10 En% carbohydrates
  Interventions: Other: diet
- high carbohydrate diet (Experimental): more than 50 En%carbohydrates
  Interventions: Other: diet

INTERVENTIONS:
Other: diet — low carbohydrate diet (< 10 EN% carbs) vs high carbohydrate diet (>50 EN% carbs)

SUMMARY:
comparing the exercise induced immune response after two weeks on a low carbohydrate (ketogenic) diet with the response after two weeks on a high carbohydrate diet.

DETAILED DESCRIPTION:
A cross-over intervention study, with a total duration of 6 weeks. An athlete follows a high, or low carbohydrate (ketogenic) diet. After 2 days a test day takes place where the athlete performs an exercise test and blood samples are taken at different time points. After that, the athlete continues following the diet for another 12 days, after which he comes back again for another identical test day. Then a 2 weeks wash-out period. After that, the athlete follows the same protocol but then with either the low (ketogenic), or high carbohydrate diet.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age: 18 - 45 y
* BMI: 18.5 - 25 kg/m2
* Hb ≥ 8.5 mmol/L, determined with blood sample from finger tip
* Minimal of 3 hours of training per week, and a maximum of 10 hours
* DKTP (diphtheria, pertussis, tetanus and polio) vaccinated (for stimulation of isolated cells (PBMC's) with tetanus toxoid)
* No asthma medication and/or anti-inflammatory medication
* No use of immunosuppressive medication
* No flu and/or travel vaccinations in the 4 months before and during the study
* Able to be present and participate at all test days
* Willing and able to follow prescribed 2 times a diet for 2 weeks in a row

Exclusion Criteria:

* Chronic illness
* Food allergies (e.g. nuts, gluten, avocado)
* Vegetarian diet
* Blood donations during study or in the 2 months prior to the study
* Use of immunosuppressive medication
* Flu and/or travel vaccination 4 months before and during the study
* Hb < 8.5 mmol/L
* Working at "Human Nutrition" - Wageningen University

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
PBMC cell differentiation changes in % | after 2 days and 2 weeks of adapted diet
  blood samples will be collected before and after exercise, the % of T-cells, NK-T-cells, B-cells, Monocytes in blood will be estimated with flow cytometrie.

SECONDARY OUTCOMES:
stress hormone Cortisol | after 2 days and 2 weeks of adapted diet
  blood samples will be collected before and after exercise, the level of cortisol will be estimated in these blood samples
ketone bodies | after 2 days and 2 weeks of adapted diet
  in urine will be detected with KetoStix
Free fatty acids | after 2 days and 2 weeks of adapted diet
  in blood will be detected with an ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mensink, Dr, Study Director — Wageningen University and Research
Locations (2):
- Netherlands (2):
  - Division of Human Nutrition, Wageningen University, Wageningen, Gelderland
  - Wageningen University and research, Wageningen, Gelderland

IPD SHARING:
Plan to Share IPD: No